CLINICAL TRIAL: NCT05001269
Title: A Phase 2 Open-Label Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Nedosiran in Pediatric Patients From Birth to 11Years of Age With Primary Hyperoxaluria and Relatively Intact Renal Function
Brief Title: Nedosiran in Pediatric Patients From Birth to 11 Years of Age With PH and Relatively Intact Renal Function
Acronym: PHYOX8
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCR-PHXC-203
Record Dates: First submitted 2021-06-30; First posted 2021-08-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Primary Hyperoxaluria; Primary Hyperoxaluria Type 1; Primary Hyperoxaluria Type 2; Primary Hyperoxaluria Type 3
Keywords: PH1; PH2; PH3; pediatric
MeSH Terms: conditions — Hyperoxaluria, Primary; Primary hyperoxaluria type 1; Primary hyperoxaluria type 2 | interventions — nedosiran

STUDY DESIGN:
Intervention Model Description: Children 2-11 years of age will begin enrolling prior to the under 2 year old age group's open.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label DCR-PHXC (Experimental): Open-Label monthly subcutaneous injection of DCR-PHXC based on age and weight.
  Interventions: Drug: nedosiran

INTERVENTIONS:
Drug: nedosiran — Monthly subcutaneous dosing throughout study period
  Other Names: DCR-PHXC

SUMMARY:
The aim of this study is to evaluate nedosiran in participants 11 years of age and younger who have Primary Hyperoxaluria with relatively intact renal function.

DETAILED DESCRIPTION:
This is an open-label, repeat-dose, Phase 2 study of nedosiran in participants 11 years of age or younger who have PH1, PH2 or PH 3 and relatively intact renal function.

Following the up-to-35- day screening period, participants will return to the clinic for monthly dosing visits through Day 180.

The total duration of this study is approximately 15 months from first participant, first visit, until last participant, last visit.

ELIGIBILITY:
Inclusion Criteria:

1. Birth to 11 years of age inclusive, at the time of signing the informed consent.
2. Documented diagnosis of PH1 or PH2 or PH3 confirmed by genotyping (historically available genotype information is acceptable for study eligibility).
3. Average spot Uox to creatinine ratio at Screening above 2 times the 95th percentile for age (Matos et al, 1999):

   * > 0.44 mol/mol in participants < 6 months
   * > 0.34 mol/mol in participants from 6 months to < 12 months
   * > 0.26 mol/mol in participants 12 months to < 2 years
   * > 0.20 mol/mol in participants from 2 to < 3 years and
   * > 0.16 mol/mol in participants from 3 to < 5 years > 0.14 mol/mol in participants from 5 to <7 years > 0.12 mol/mol in participants from 7 to 11 years
4. Estimated GFR at Screening ≥ 30 mL/min normalized to 1.73 m2 BSA. See Section 8.2.6.1 for equations. For infants aged less than 12 months, serum creatinine below the 97th percentile of a healthy population (Boer et al., 2010).
5. Participants must have been on a stable treatment regimen for PH for 3 months prior to Day 1 and parent(s)/legal guardian should be willing to ensure participant remains on the same stable treatment regimen during the study. Dose adjustments for interval weight gain are acceptable.
6. Male or Female

   Male participants:

   A male participant with a female partner of childbearing potential must agree to use contraception, as detailed in Section 10.5.2, during the treatment period and for at least 12 weeks after the last dose of study intervention and refrain from donating sperm during this period.

   Female participants:

   A female participant is eligible to participate if she is not pregnant (see Section 10.5.1), not breastfeeding, and at least 1 of the following conditions applies:

   Not a woman of childbearing potential (WOCBP) as defined in Section 10.5.1 OR A WOCBP who agrees to follow the contraceptive guidance in Section 10.5.2 during the treatment period and for at least 12 weeks after the last dose of study intervention.

   Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Note: If the childbearing potential changes after start of the study (e.g., a premenarchal female participant experiences menarche) or the risk of pregnancy changes (e.g., a female participant who is not heterosexually active becomes active), the participant must discuss this with the Investigator, who should determine if a female participant must begin a highly effective method of contraception or a male participant must use a condom. If reproductive status is questionable, additional evaluation should be considered.
7. Participant's parent or legal guardian is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

   a. For children younger than 12 years of age, assent will be based on local regulation. If assent is required, participant must be able to provide written assent for participation.
8. A legal guardian or primary caregiver must be available to help the study-site personnel ensure follow up; accompany the participant to the study site on each assessment day according to the SoA (e.g., able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures); consistently and consecutively be available to provide information on the participant using the rating scales during the scheduled study visits; accurately and reliably dispense study intervention as directed.
9. Affiliated with or is a beneficiary of a health insurance system (if applicable per national regulations)

Exclusion Criteria:

1. Prior renal or hepatic transplantation; or planned transplantation within the study period
2. Currently receiving dialysis or anticipating requirement for dialysis during the study period
3. Plasma oxalate (Pox) > 30 μmol/L at Screening
4. Documented evidence of clinical manifestations of severe systemic oxalosis (including preexisting retinal, heart, or skin calcifications, or history of severe bone pain, pathological fractures, or bone deformations)
5. Presence of any condition or comorbidities that would interfere with study compliance or data interpretation or potentially impact participant's safety including, but not restricted to:

   1. Severe intercurrent illness
   2. Known causes of active liver disease/injury or transaminase elevation (e.g., alcoholic liver disease, nonalcoholic fatty liver disease/steatohepatitis [NAFLD/NASH])
   3. History of serious mental illness that includes, but is not limited to, schizophrenia, bipolar disorder, or severe depression requiring hospitalization or pharmacological intervention
   4. Clinically relevant history or presence of cardiovascular, respiratory, gastrointestinal, hematological, lymphatic, neurological, musculoskeletal, genitourinary, immunological diseases, including dermatological including rash, severe eczema or dermatitis, or connective tissue diseases or disorders
6. Use of an RNAi drug within the last 6 months
7. History of 1 or more of the following reactions to an oligonucleotide-based therapy:

   1. Severe thrombocytopenia (platelet count ≤ 100,000/µL)
   2. Hepatotoxicity, defined as ALT or AST > 3 times the upper ULN and total bilirubin > 2 × ULN or INR > 1.5
   3. Severe flu-like symptoms leading to discontinuation of therapy
   4. Localized skin reaction from the injection (graded severe) leading to discontinuation of therapy
   5. Coagulopathy/clinically significant prolongation of clotting time
8. Participation in any clinical study in which they received an IMP within 4 months or 5 times the half-life of the drug (whichever is longer) before Screening

   a. For IMPs with the potential to reduce urine and/or plasma oxalate concentrations, these concentrations must have returned to historical baseline levels prior to Screening
9. Liver function test (LFT) abnormalities: ALT and/or AST > 1.5 × ULN for age and gender
10. Known hypersensitivity to nedosiran, or any of its ingredients
11. Inability or unwillingness to comply with the specified study procedures, including the lifestyle considerations detailed in Section 5.3.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Efficacy: Percent change in urinary oxalate to creatinine ratio | 180 days
  Evaluate the effect of nedosiran on percent change in urinary oxalate-to-creatinine ratio
Efficacy: Absolute change in urinary oxalate to creatinine ratio | 180 days
  Evaluate the effect of nedosiran on absolute change in urinary oxalate-to-creatinine ratio

SECONDARY OUTCOMES:
Safety: Incidence of Events | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger based on treatment emergent adverse events, and serious adverse events.
Safety: Changes from baseline in ECG: Rhythm | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in ECG.
Safety: Changes from baseline in ECG: Ventricular Rate | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in ECG.
Safety: Changes from baseline in ECG: PR interval | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in ECG.
Safety: Changes from baseline in ECG: QRS duration | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in ECG.
Safety: Changes from baseline in ECG: QT interval | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in ECG.
Safety: Changes from baseline: Physical Exam | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in physical exam and physician review of systems based on CTCAE v5.0
Safety: Changes from baseline in Vitals: temperature | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in vital signs.
Safety: Changes from baseline in Vitals: pulse rate | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in vital signs.
Safety: Changes from baseline in Vitals: respiratory rate | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in vital signs.
Safety: Changes from baseline in Vitals: blood pressure | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in vital signs.
Safety: Changes from baseline: Labs - Hematology | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Clinical Chemistry | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Coagulation | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Antibody | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Plasma Oxalate | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Urinalysis | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
Safety: Changes from baseline: Labs - Urine Oxalate | 180 days
  Characterize the safety of nedosiran in children 11 years of age and younger changes from baseline in clinical laboratory tests.
To characterize the PK of DCR PHXC in patients with PH by observing secondary parameters of the area under the curve. | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including secondary parameters of area under the curve (AUC)
To characterize the PK of DCR PHXC in patients with PH by observing maximum observed concentration (Cmax). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including maximum observed concentration (Cmax)
To characterize the PK of DCR PHXC in patients with PH by observing minimum concentration (Cmin). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including minimum observed concentration (Cmin)
To characterize the PK of DCR PHXC in patients with PH by observing maximum concentration (Tmax). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including time to maximum concentration (Tmax)
To characterize the PK of DCR PHXC in patients with PH by observing terminal elimination half-life (t1/2). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including terminal elimination half-life (t1/2)
Efficacy: eGFR changes | 180 days
  Evaluate the effect of nedosiran on eGFR from baseline

OTHER OUTCOMES:
Change from Baseline in Plasma Oxalate Concentration | 180 days
  Assess the effect of DCR-PHXC on Plasma Oxalate concentration from baseline
Change from Baseline number of kidney stones | 180 days
  Assess the effect of DCR-PHXC on stone burden from baseline on annualized stone events
Change from baseline PedsQL™ | 180 days
  Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL™)
Change from baseline WPAI | 180 days
  Change from Baseline in the Work Productivity and Activity Impairment Questionnaire: Primary Hyperoxaluria V2.0, Clinical Practice Version (WPAI:PH, V2.0, CPV) - Caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Sarb Shergill, PhD, Study Director — Dicerna Pharmaceuticals, Inc., a Novo Nordisk company
Locations (13):
- Clinical Research Site, Rochester, Minnesota, United States
- Clinical Research Site, Hamilton, Ontario, Canada
- Germany (2):
  - Clinical Trial Site, Bonn
  - Clinical Research Site, Heidelberg
- Clinical Trial Site, Roma, Italy
- Japan (2):
  - Clinical Research Site, Fukuoka
  - Clinical Research Site, Nagoya
- Clinical Research Site, Beirut, Lebanon
- Clinical Research Site, Bialystok, Poland
- Clinical Research Site, Barcelona, Spain
- Clinical Research Site, Yenimahalle, Ankara, Turkey (Türkiye)
- Clinical Trial Site, Dubai, United Arab Emirates
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang S, Gamallo P, Rawson V. Population Pharmacokinetic and Pharmacodynamic Modelling and Simulation for Nedosiran Clinical Development and Dose Guidance in Pediatric Patients with Primary Hyperoxaluria Type 1. Clin Pharmacokinet. 2025 Sep;64(9):1395-1411. doi: 10.1007/s40262-025-01540-1. Epub 2025 Jul 2. PMID 40601241
- [Derived] Cox JH, Boily MO, Caron A, Sheng T, Wu J, Ding J, Gaudreault S, Chong O, Surendradoss J, Gomez R, Lester J, Dumais V, Li X, Gumpena R, Hall MD, Waterson AG, Stott G, Flint AJ, Moore WJ, Lowther WT, Knight J, Percival MD, Tong V, Oballa R, Powell DA, King AJ. Characterization of CHK-336, A First-in-Class, Liver-Targeted, Small-Molecule Lactate Dehydrogenase Inhibitor for Hyperoxaluria Treatment. J Am Soc Nephrol. 2025 Apr 7;36(8):1535-1547. doi: 10.1681/ASN.0000000690. PMID 40193200